CLINICAL TRIAL: NCT07181902
Title: Postoperative Recovery Quality After Cesarean Section: Comparing Erector Spinae and Retrolaminar Blocks Using Turkish Version of the Obstetric Quality-of-Recovery Score (ObsQoR-11T) in a Turkish Cohort
Brief Title: Postoperative Recovery Quality After Cesarean Section: Comparing Erector Spinae and Retrolaminar Blocks Using Turkish Version of the Obstetric Quality-of-Recovery Score in a Turkish Cohort (ObsQoR-11T)
Status: Not yet recruiting | Type: Observational
Sponsor: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Responsible Party: Principal Investigator, Serpil Bayındır, Specialist Physician, Elazıg Fethi Sekin Sehir Hastanesi
Other Study IDs: FSCH-SB-2024/09CSRLB
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pain Management
Keywords: Cesarean Section; Retrolaminar Block; ObsQoR-11T; Erector Spinae Plane Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESP Group - Erector Spinae Plane Block: Patients receiving ultrasound-guided Erector Spinae Plane (ESP) block immediately after cesarean section under spinal anesthesia. The block is performed at T9 level using 20 mL of 0.25% bupivacaine. Standard perioperative care and analgesia protocols are applied to all participants. Postoperative recovery quality, pain scores, opioid consumption, and adverse events are recorded.
  Interventions: Procedure: Erector Spinae Plane Block (ESP)
- RLB Group - Retrolaminar Block: Patients receiving ultrasound-guided Retrolaminar Block (RLB) immediately after cesarean section under spinal anesthesia. The block is performed at T9 level using 20 mL of 0.25% bupivacaine. Standard perioperative care and analgesia protocols are applied. Postoperative recovery quality, pain scores, opioid consumption, and adverse events are recorded.
  Interventions: Procedure: Retrolaminar Block (RLB)

INTERVENTIONS:
Procedure: Erector Spinae Plane Block (ESP) — Ultrasound-guided ESP block performed immediately after cesarean section at T9 level using 20 mL of 0.25% bupivacaine. Standard perioperative care and analgesia protocols are applied.
  Groups: ESP Group - Erector Spinae Plane Block
Procedure: Retrolaminar Block (RLB) — Ultrasound-guided Retrolaminar Block performed immediately after cesarean section at T9 level using 20 mL of 0.25% bupivacaine. Standard perioperative care and analgesia protocols are applied.
  Groups: RLB Group - Retrolaminar Block

SUMMARY:
Study Design This retrospective observational study aims to evaluate and compare the effects of two regional anesthesia techniques, Erector Spinae Plane (ESP) block and Retrolaminar Block (RLB), on postoperative recovery quality in women undergoing elective cesarean section (CS). Postoperative pain after CS is common, particularly in the first 24-72 hours, and can affect mobility, breastfeeding, and overall well-being. Effective pain management is therefore critical for both patient comfort and maternal-infant bonding.

Participants and Methods Medical records of adult women aged 18-45 years, with a singleton pregnancy at ≥37 weeks, who underwent elective CS under spinal anesthesia in our clinic, were retrospectively reviewed. Patients who had received either ESP or RLB immediately after surgery were included. Both blocks had been performed under ultrasound guidance at the T9 level using 20 mL of 0.25% bupivacaine, according to institutional practice. Standard perioperative care and analgesia protocols were applied to all patients.

Outcomes The primary outcome was postoperative recovery quality, assessed 24 hours after surgery using the Turkish version of the Obstetric Quality-of-Recovery Score (ObsQoR-11T), a validated tool addressing physical, emotional, and functional aspects of recovery. Secondary outcomes included postoperative pain intensity (Visual Analog Scale), opioid consumption, adverse events, and patient satisfaction, as documented in patient files.

Conclusion This retrospective study will provide evidence on which block technique more effectively improves recovery quality after CS and may help optimize postoperative analgesia strategies in Turkish obstetric populations.

DETAILED DESCRIPTION:
METHODS 1.1. Study Design and Settings

This was a retrospective, single-center observational study conducted to evaluate the effects of ESP and RLB on postoperative pain, opioid consumption, and patient satisfaction in women undergoing cesarean section. The study was carried out at Elazığ Fethi Sekin City Hospital, a tertiary care center in Elazığ, Türkiye. Medical records of eligible patients were reviewed for the analysis. The study protocol was approved by the local institutional ethics committee and conducted in accordance with the principles of the Declaration of Helsinki.

1.2. Participants

The study population consisted of adult women who had undergone elective CS at Elazığ Fethi Sekin City Hospital between [start date] and [end date].

Inclusion Criteria

Women aged 18-45 years who underwent elective CS under spinal anesthesia.

Gestational age ≥37 weeks, singleton pregnancy.

Received either ESP or RLB for postoperative analgesia, documented in anesthesia records.

ASA Physical Status II-III.

Completion of ObsQoR-11T questionnaire at 24 hours postoperatively.

Exclusion Criteria

Emergency cesarean delivery.

Multiple pregnancy or preterm delivery (<37 weeks).

Severe maternal or obstetric complications (e.g., preeclampsia, placenta previa, placenta accreta spectrum).

BMI ≥40 kg/m².

Significant systemic disease (e.g., severe cardiac, respiratory, renal, or hepatic disease).

Fetal or placental anomalies.

History of chronic pain syndromes, opioid dependence, or long-term analgesic use.

Neurological, psychiatric, or cognitive disorders interfering with pain perception or questionnaire completion.

Missing or incomplete data in the medical records.

1.3. Protocol and Outcome Measures

Anesthesia and Postoperative Analgesia All patients had received a standardized spinal anesthesia protocol. During surgery, patients had been positioned supine with a 15° left tilt and given oxygen at 4 L/min via face mask. Adequate sensory block at the T4-T6 level had been confirmed before the CS procedure began.

Approximately 30 minutes before the end of surgery, intravenous 1 g paracetamol and 50 mg dexketoprofen had been administered as part of multimodal postoperative analgesia. Before recovery, ESP or RLB was performed at the T9 level under ultrasound guidance.

Patients were classified into two groups according to the block technique documented in anesthesia charts:

ESP Group: Bilateral ESP block at T9 with 20 mL of 0.25% bupivacaine per side.

RLB Group: Bilateral RLB at T9 with 20 mL of 0.25% bupivacaine per side.

All blocks had been performed by experienced anesthesiologists trained in ultrasound-guided techniques. Postoperatively, patients were monitored in the recovery unit and transferred to the postpartum ward once stable (Modified Aldrete score ≥9).

Surgical Technique Only patients whose records documented a standardized surgical technique were included. All elective CS operations had been performed using a Pfannenstiel skin incision and a lower-segment transverse uterine incision. Uterine closure had been performed with a single layer of absorbable sutures.

Primary Outcome The primary outcome was postoperative recovery quality, assessed at 24 hours using the ObsQoR-11T score recorded in patient files.

Secondary Outcomes

Demographic and clinical characteristics (age, BMI, ASA status, comorbidities, obstetric history).

Intraoperative data: duration of surgery and anesthesia.

Postoperative analgesic requirements: time to first rescue analgesic, total analgesic consumption within 24 hours.

Pain intensity (VAS at rest and on coughing at 1, 6, 12, and 24 hours).

Adverse events (nausea, vomiting, hypotension, bradycardia, block-related complications).

Patient satisfaction scores as documented in follow-up notes.

1.4. Sample Size

As this was a retrospective study, no prior sample size calculation was performed. All patients who met the inclusion criteria during the study period were included in the analysis.

ELIGIBILITY:
Inclusion Criteria

* Women aged 18-45 years, scheduled for elective cesarean delivery under spinal anesthesia.
* Gestational age ≥37 weeks, singleton pregnancy.
* Undergoing either ESP or RLB for postoperative analgesia.
* ASA Physical Status II-III.
* Ability to understand and complete ObsQoR-11T questionnaire.
* Provided written informed consent prior to participation. Exclusion Criteria
* Emergency cesarean delivery.
* Multiple pregnancy, preterm delivery (<37 weeks),
* Severe maternal or obstetric complications (e.g., preeclampsia, placenta previa, placenta accreta spectrum), regardless of urgency.
* BMI ≥40 kg/m²
* Significant systemic diseases (e.g., severe cardiac, respiratory, renal, or hepatic disease).
* Fetal or placental anomalies.
* History of chronic pain syndromes, opioid dependence, or long-term analgesic use.
* Neurological, psychiatric, or cognitive disorders that may interfere with pain perception or questionnaire completion.
* Patients who declined participation or did not provide informed consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study includes adult women undergoing elective cesarean section at Elazığ Fethi Sekin City Hospital. Participants will receive either an Erector Spinae Plane (ESP) block or a Retrolaminar Block (RLB) for postoperative analgesia and will be followed for postoperative recovery quality and pain outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative Recovery Quality After Cesarean Section (ObsQoR-11T) | 24 hours postoperatively
  The primary outcome is the quality of postoperative recovery, assessed using the Turkish version of the Obstetric Quality-of-Recovery Score (ObsQoR-11T). This validated questionnaire evaluates multidimensional aspects of recovery, including patient comfort, physical and emotional well-being, and functional status. Scores are recorded 24 hours after cesarean section to compare recovery between ESP and RLB groups.

SECONDARY OUTCOMES:
Postoperative Pain Intensity (Visual Analog Scale) | 1, 6, 12, and 24 hours postoperatively
  Pain intensity at rest and during coughing is assessed using the Visual Analog Scale (VAS; 0 = no pain, 10 = worst imaginable pain) at 1, 6, 12, and 24 hours postoperatively in both ESP and RLB groups.
Total Analgesic Consumption | 0-24 hours postoperatively
  Total postoperative analgesic consumption, including opioids and non-opioid medications, is recorded during the first 24 hours after cesarean section to compare ESP and RLB groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Elazığ Fethi Sekin City Hospital, Elâzığ, Seçiniz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided